CLINICAL TRIAL: NCT00112099
Title: Randomized Controlled Trial to Evaluate Splenectomy in Total Gastrectomy for Proximal Gastric Carcinoma: JCOG0110
Brief Title: GCSSG-SPNX: Trial to Evaluate Splenectomy in Total Gastrectomy for Proximal Gastric Carcinoma: JCOG0110
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG 0110; C000000004
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Neoplasm
Keywords: gastric neoplasm; gastrectomy; splenectomy; randomized trial; T2, T3 and T4 carcinoma in the proximal third of the stomach
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: Surgery: Splenectomy
  Interventions: Procedure: Surgery: Splenectomy
- 2 (Experimental): Procedure/Surgery: Surgery: Spleen-preservation
  Interventions: Procedure: Surgery: Spleen-preservation

INTERVENTIONS:
Procedure: Surgery: Splenectomy — Procedure/Surgery: Surgery: Splenectomy
  Arms: 1
Procedure: Surgery: Spleen-preservation — Procedure/Surgery: Surgery: Spleen-preservation
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the role of splenectomy in potentially curative total gastrectomy for proximal gastric carcinoma in terms of survival benefit and post-operative morbidity.

DETAILED DESCRIPTION:
European clinical trials of gastrectomy showed that splenectomy is an important risk factor for post-operative morbidity and mortality. Retrospective comparisons suggested that splenectomy is associated with poor long term survival. However, Japanese studies revealed that 20 - 30 % of patients with non-early carcinoma in the proximal stomach have nodal metastasis in the splenic hilum and therefore, pancreas-preserving splenectomy is part of the standard operation in specialized centers where splenectomy is not considered a risk factor for operative mortality. There have been no prospective randomized trials to evaluate the survival benefit of splenectomy in total gastrectomy for proximal gastric cancer.

Comparison: Total gastrectomy with pancreas-preserving splenectomy versus total gastrectomy without splenectomy

ELIGIBILITY:
Inclusion Criteria:

Preoperatively

* Histologically proven adenocarcinoma
* T2 or deeper lesion in the upper third of the stomach without involvement of the greater curvature or esophageal invasion, irrespective of the primary tumor location or existence of multiple foci
* No distant metastasis, not linitis plastica ('Borrmann 4'), not stump carcinoma, no prior treatment for 364 Randomized trial for splenectomy gastric cancer
* Sufficient organ function
* Written informed consent.

Intra-operatively

* T2/T3/T4 and N0/N1/N2, no tumor on the greater curvature, no direct invasion of the pancreas or spleen, negative peritoneal lavage cytology
* No apparent nodal metastasis in the splenic hilum or along the splenic artery

Exclusion Criteria:

* Liver cirrhosis or portal hypertension
* Idiopathic thrombocytopenic purpura
* Severe pulmonary dysfunction
* Synchronous or metachronous (within 5 years) malignancy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2002-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | During the study conduct

SECONDARY OUTCOMES:
Post-operative morbidity | 5 years
operation time | day of the operation
perioperative blood loss | 3 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Sasako, MD, PhD, Study Chair — Hyogo Medical University
Locations (35):
- Japan (35):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Fujita Health University, Toyoake,Kutsukake-cho,Dengakugakubo,1-98, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Gifu Municipal Hospital, Gifu,Kashima-cho,7-1, Gifu
  - Hiroshima City Hospital, Hiroshima,Naka-ku,Motomachi,7-33, Hiroshima
  - Itami City Hospital, Itami,Koyaike,1-100, Hyōgo
  - Iwate Medical University, Morioka,Uchimaru,19-1, Iwate
  - Kagoshima University,Faculty of Medicine, Kagoshima,Sakuragaoka,8-35-1, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Kyoto Second Red Cross Hospital, Kyoto,Kamigyo-ku,Kamanza-Marutamachi,355-5, Kyoto
  - Miyagi Cancer Center, Natori,Medeshima-Shiode,Nodayama,47-1, Miyagi
  - National Hospital Organization, Sendai Medical Center, Sendai,Miyagino-ku,Miyagino,2-8-8, Miyagi
  - Nagaoka Chuo General Hospital, Nagaoka,Kawasaki,2041, Niigata
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Tsubame Rosai Hospital, Tsubame,Sawatari,633, Niigata
  - Oita University Fuculty of Medicine, Oita1-1,Hasama-machi,Oogaoka, Oita Prefecture
  - Osaka National Hospital, Osaka,Chuo-ku,Hoenzaka,2-1-14, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - Sakai Municipal Hospital, Sakai,Minamiyasuicho,1-1-1, Osaka
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Toyonaka Municipal Hospital, Toyonaka,Shibaharacho,4-14-1, Osaka
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - National Defense Medical College, Tokorozawa,Namiki,3-2, Saitama
  - Shizuoka General Hospital, Shizuoka,Aoi-ku,Kitaando,4-27-1, Shizuoka
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku,Honkomagome,3-18-22, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - International Medical Center of Japan, Shinjuku-ku,Toyama,1-21-1, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku,Koutoubashi,4-23-15, Tokyo
  - Toyama Prefectural Central Hospital, Toyama,Nishinagae,2-2-78, Toyama
  - Wakayama Medical University, School of Medicine, Wakayama,Kimiidera,811-1, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- [Background] Sano T, Yamamoto S, Sasako M; Japan Clinical Oncology Group Study LCOG 0110-MF. Randomized controlled trial to evaluate splenectomy in total gastrectomy for proximal gastric carcinoma: Japan clinical oncology group study JCOG 0110-MF. Jpn J Clin Oncol. 2002 Sep;32(9):363-4. doi: 10.1093/jjco/hyf085. PMID 12417603
- See also: Related Info — http://www.jcog.jp/